CLINICAL TRIAL: NCT00210873
Title: An Open-label Study of the Safety and Efficacy of Topiramate for the Prophylaxis of Chronic Migraine: Extension Study to CAPSS-276
Brief Title: An Open Label Extension of a Study of Topiramate in Chronic Migraine.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Collaborators: Ortho-McNeil Neurologics, Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CR004672
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2011-06-10 (Estimated); Status verified 2010-05

CONDITIONS: Migraine
Keywords: Migraine; headache; chronic; prevention
MeSH Terms: conditions — Migraine Disorders; Headache; Bronchiolitis Obliterans Syndrome | interventions — Topiramate

INTERVENTIONS:
Drug: topiramate

SUMMARY:
The purpose of this study is to assess the long-term safety and effectiveness of topiramate for the prevention of headaches in adults with chronic migraine. Topiramate has been approved to prevent migraine headaches.

DETAILED DESCRIPTION:
Migraine headaches can be disabling and can interfere with work and a person's quality of life. Preventing these headaches before they start is the best option. Topiramate, an anti-seizure medication, has been shown to help prevent migraine headaches from occurring. This is an open-label study that is an extension of a previous study (CAPSS-276) of Topiramate in chronic migraine. It includes patients who completed the previous study or who stopped the study early after taking study drug for at least 4 weeks of maintenance treatment due to lack of efficacy. The current study will involve a 4-week Blinded Transition Phase during which patients will be titrated up to a daily topiramate dose of 100 milligrams (or the maximum tolerated dose, whichever is less). Then there will be a 12-week Open-Label Maintenance Phase during which the topiramate dose may be adjusted according to effectiveness and tolerance, but not to exceed a daily dose of 400 milligrams. After this period, patients will be tapered off topiramate (Taper/Exit Phase). The length of the taper/exit phase may vary based on the dose the patient was taking during the open label maintenance phase. While on topiramate, patients will record daily entries in their headache records. Patients will also be asked questions to help assess their quality of life. Both patients and doctors will be asked questions at the end of the study about their impressions of change with respect to the patient's migraine headaches. Patients will also have physical and neurological examinations and laboratory tests performed during the study. The objective of this study is to evaluate the long-term safety and effectiveness of topiramate for the prevention of chronic migraine headaches. Topiramate oral tablets, 25 milligrams per tablet, will be given in the morning and evening to a dose not to exceed 400 milligrams per day or to the maximum tolerated dose, whichever is less

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of chronic migraine
* successfully finished double-blind portion of the CAPSS-276 study or discontinued the study after a minimum of 4 weeks maintenance treatment due to lack of effect of study drug
* in generally good health
* able to take medicine orally
* if female, using birth control.

Exclusion Criteria:

* Cannot have a more painful condition than the headache pain
* cannot be taking any other medications not allowed by the study protocol
* no abnormal liver tests
* not compliant with study medication during the CAPSS-276 study
* cannot be pregnant or breast-feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2004-02; Study Completion 2005-08 (Actual)

PRIMARY OUTCOMES:
Patient diaries for number & severity of migraine or migrainous headaches, symptoms, & other medications used; Migraine Disability Assessment, Migraine-Specific Quality of Life, Physicians & Subjects Global Impression of Change for quality of life

SECONDARY OUTCOMES:
Adverse event reports; physical examinations; vital signs; laboratory tests for safety

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- See also: An open label extension of a study of Topiramate in chronic migraine. — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=619&filename=CR004672_CSR.pdf